CLINICAL TRIAL: NCT01974778
Title: A Role for Brown Adipose Tissue in Postprandial Thermogenesis?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant numbers too low. Could not ingest required fat.
Sponsor: Bayside Health (Other Government)
Responsible Party: Principal Investigator, Ms. Rowan Frew, Ms, Bayside Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 345-13
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Meal
  Interventions: Dietary Supplement: Meal
- Control (Placebo Comparator): Water
  Interventions: Dietary Supplement: Meal

INTERVENTIONS:
Dietary Supplement: Meal — Meal

SUMMARY:
Brown adipose (fat) tissue (BAT) is a type of fat tissue found in certain small rodents and human babies that is capable of extremely high rates of energy burning. We now know that in adult humans it is present and also able to burn energy.

In addition to increased energy expenditure during cold exposure, energy burning is also increased after consuming a meal. Animal studies have shown that part of this additional energy consumption is contributed by BAT. In the present study we will aim to examine whether BAT activity is increased after a meal.

DETAILED DESCRIPTION:
The purpose of this project is to measure whether BAT activity (during which BAT increases energy burning) increases in response to ingestion of a meal.

BAT is one of two types of fat, (the other being white fat), which is found in humans and other mammals. In this study we aim to further our understanding of how BAT works in humans. Studies in animals show that in addition to cold exposure, BAT is also activated by ingestion of a meal, and to different amounts depending on the meal composition, and more importantly, total energy content. However we have only a very limited understanding of BAT function in response to meals in humans. Since BAT function is defective in obesity, and its activity and function are impacted by diet, here we will find out whether a single high energy meal composed entirely of lipid (fat) can increase BAT activity. In future these findings and those of subsequent studies may have important implications for the management of obesity and related diseases.

A total of 20 people will participate in this project. Participation will involve a total of 3 visits, including a screening visit, 2 experimental visits consumption of the treatment meal on one visit, and the placebo (dummy) on the other in a randomised order.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 19 - 35 years
* Unmedicated for the previous 2 months
* No major illness
* BMI 17-40 kg/m2

Exclusion Criteria:

* Unable to give informed consent
* Smokers
* Participant in research projects involving ionising radiation within the past 5 years, excluding dual energy x-ray absorptiometry scans conducted in prior studies
* Claustrophobia
* Fasting plasma glucose > 6.0 mmol/L

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
BAT activity | 2 years
  Analysis of PET/CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn Kingwell, Professor, Principal Investigator — Baker IDI Heart & Diabetes Institute
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia